CLINICAL TRIAL: NCT03996512
Title: Early Active Controlled Motion (EACM) Rehabilitation Protocol Post Open Reduction and Internal Fixation (ORIF) of Scaphoid Fractures: A Pilot Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment issues. Inclusion Criteria was strict due to the experimental nature of intervention
Sponsor: University of Florida (Other)
Collaborators: Performance Health (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB201900006
Record Dates: First submitted 2019-06-21; First posted 2019-06-24 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Scaphoid Fixation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post scaphoid fracture with screw fixation (Experimental): Post surgical rehabilitation using an early active controlled wrist motion rehab protocol that limits the amount of proximal carpal row loading forces
  Interventions: Other: Early Active Controlled Motion (EACM)

INTERVENTIONS:
Other: Early Active Controlled Motion (EACM) — Early active controlled wrist motion rehab protocol using that will allow midcarpal row motion.

SUMMARY:
There is poor research supporting the benefits of Early Active Controlled Motion (EACM) protocols post operative scaphoid fixation. Advances in surgical fixation technique for scaphoid fractures should allow for start of earlier mobilization, however there is little evidence in the literature that supports the use of these protocols within the early phases of healing. The study uses a pre-experimental design with purposeful sample population recruitment.

ELIGIBILITY:
Inclusion Criteria:

* Date of injury and diagnosis: scaphoid fracture less than 3 weeks old
* Waist fractures in the middle 1/3 and distal pole 1/3 of scaphoid bone.
* Surgical procedure includes ORIF with screw fixation and/or percutaneous pin with screw fixation.
* To be included in the study the patient needs to have started rehab within the first 10 days after surgery date.

Exclusion Criteria:

* Proximal pole scaphoid fracture
* Past medical history of diabetes and other peripheral vascular disorders.
* History of osteopenia and osteoporosis.
* Previously failed ORIF of scaphoid
* Neurovascular or nerve lesion to the involved upper extremity
* Cognitive deficits related to memory, attention span, judgment as documented in the EMR or need for a legal guardian to be a medical proxy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-01-19 (Actual); Study Completion 2021-01-19 (Actual)

PRIMARY OUTCOMES:
functional outcome range of motion | at entry and up to 12 months
  Using a goniometer measuring the angle of wrist flexion and extension
  NEED TO ENTER EXPECTED ROM ranges

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Mersch, Principal Investigator — University of Florida

IPD SHARING:
Plan to Share IPD: No